CLINICAL TRIAL: NCT04025099
Title: Internal Cues Versus External Cues for Eating and Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Carly R Pacanowski, Principal Investigator, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1408101
Record Dates: First submitted 2019-07-12; First posted 2019-07-18 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Eating Behavior; Body Image; Diet Habit; Dietary Habits
Keywords: intuitive eating; body positive yoga; weight management; cardiovascular fitness; interoceptive awareness; embodiment; internal cues; external cues
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This three-armed randomized, controlled trial will assess the effects of a novel internal cues intervention (treatment group; intuitive eating and body positive yoga) compared to an active control group consisting of traditional healthy weight sessions, following standardized government recommendations for eating and activity, and a no-treatment control group completing assessments only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internal Cues (Experimental): Over 10 weeks, participants will be asked to participate in the following:
  1. Classes (held in STAR Tower 419/420 IPE Space and Conference Room 413)
     * One ~60-minute Intuitive Eating class per week (total = 10 classes);
     * Two ~60-minute yoga classes per week (total = 20 classes);
     * Repeat one of the ~60-minute yoga classes each week on the participants' own, in a space participants feel comfortable, using a video recording (total = 10 classes).
  2. Assessments (held in STAR tower)
     * Three ~60-minute assessments* which will include:
       1. Height & weight measurements (taken privately)
       2. A questionnaire that asks about participants' relationship with their body and eating and activity behaviors
       3. Collection of participants' heart rate overnight (on their own)
       4. Collection of participants' saliva three times in one day (on their own)
  Interventions: Other: Internal Cues
- External Cues (Active Comparator): Over the next 10 weeks, participants will be asked to participate in the following:
  1. Classes (held in STAR Tower 419/420 IPE Space)
     * One ~60-minute Healthy Eating class per week (total = 10 classes);
     * Participants will be provided with a UD group fitness membership. Using this membership, participants will be asked to attend at least 2 cardio fitness classes per week and do an additional 30 minutes of heart-raising activity on participants' own (total = 3 exercise sessions/week).
  2. Assessments (held in STAR tower)
     * Three ~60-minute assessments* which will include:
       1. Height & weight measurements (taken privately)
       2. A questionnaire that asks about participants' relationship with their body and eating and activity behaviors
       3. Collection of participants' heart rate overnight (on their own)
       4. Collection of participants' saliva three times in one day (on their own)
  Interventions: Other: External Cues
- Assessment Only (No Intervention): Over the next 10 weeks, participants will be asked to participate in the following:
  a. Assessments (held in STAR tower)
  •Three ~60-minute assessments* which will include:
  1. Height & weight measurements (taken privately)
  2. A questionnaire that asks about participants' relationship with their body and eating and activity behaviors
  3. Collection of participants' heart rate overnight (on their own)
  4. Collection of participants' saliva three times in one day (on their own)

INTERVENTIONS:
Other: Internal Cues — The intuitive eating curriculum that was pilot tested and adapted has been modified for use for the Internal Cues group with college-aged females for delivery over a 10-week time period.
  The classes will be delivered by two Registered Dietitians and Certified Intuitive Eating Counselors from the University of Delaware, Julia Katcher and Maryann Eastep.
  During the Internal Cues group's intuitive eating classes, participants will, as a group, eat dinner that is prepared by ServSafe certified undergraduate dietetics students in the test kitchen in the STAR Tower. This dinner will allow the participants to experientially learn the intuitive eating principles taught in class.
  The yoga classes will be adapted to all levels of experience, mobility, and body size. Specific breathing techniques and body positive language will be incorporated into a body-positive yoga training done by Ms. Lisa Jones, RYT.
  Arms: Internal Cues
Other: External Cues — The 10-week traditional healthy weight program for the External Cues group was created by a Graduate Assistant based on MyPlate principles.
  The External Cues classes will be delivered by two Registered Dietitians from the University of Delaware, Julia Katcher and Maryann Eastep.
  During the External Cues group's healthy eating classes, participants will, as a group, eat dinner that is prepared by ServSafe certified undergraduate dietetics students in the test kitchen in the STAR Tower. This dinner will allow the participants to experientially learn how to properly portion their meals to meet their caloric needs, in line with traditional education about weight control.
  Students randomized to the External Cues group will receive a UD fitness pass and will be able to choose from select cardio-based fitness classes in order to meet public health recommendations for physical activity.
  Arms: External Cues

SUMMARY:
The majority of female undergraduate students experience disordered eating and/or weight gain, increasing the risk for two serious public health problems, eating disorders and obesity. Traditional nutrition education about weight control delivered during college has not been effective and may even exacerbate these problems. Thus, the investigators propose that instead of focusing on external information as taught by nutrition education (e.g. 'calories in, calories out', quantification and cognitive processing of nutrition information), at-risk females be trained to become more attuned to their internal hunger and fullness signaling to set them on a trajectory for decreased chronic disease risk as they age.

DETAILED DESCRIPTION:
The proposed study, Internal versus External Cues for Eating and Activity, will collect data on within-person changes in psychological (e.g. attunement with bodily signals, eating and activity behaviors) and physiological (e.g., body mass index, heart rate, saliva) markers of risk for both eating disorders and obesity in female University of Delaware students. Outcomes will be assessed at baseline, mid-treatment, end-of-treatment, and one-year follow-up. This three-armed randomized, controlled trial will assess the effects of a novel internal cues intervention (treatment group; intuitive eating and body positive yoga) compared to an active control group consisting of traditional healthy weight sessions, following standardized government recommendations for eating and activity, and a no-treatment control group completing assessments only. The Internal Cues group will attend one intuitive eating session and take three body-positive yoga sessions weekly for ten weeks. The External Cues group will attend one healthy weight class and three cardiovascular-based exercise sessions each week for ten weeks. The Assessment Only no-treatment control group will only attend assessments. The curriculum for the intuitive eating classes (previously piloted and revised accordingly) and healthy weight classes (modeled off of classes offered at universities and government-available recommendations and educational documents) will be taught by two Registered Dietitians who are Certified Intuitive Eating Counselors. The yoga classes will be taught by a Registered Yoga Instructor trained in Body Positive Yoga and in a curriculum specifically designed for UD students (funded by Dean Matt). During the Internal Cues group's intuitive eating classes, participants will, as a group, eat dinner that is prepared by ServSafe certified undergraduate dietetics students in the test kitchen in the STAR Tower. This dinner will allow the participants to experientially learn the intuitive eating principles taught in class. The External Cues group will receive an identical dinner during the class period but they will learn how to properly portion their meals to meet their caloric needs, in line with traditional education about weight control. Finally, students randomized to the External Cues group will receive a UD fitness pass and will be able to choose from select cardio-based fitness classes in order to meet public health recommendations for physical activity.

Additionally, the interventionists for both the Internal Cues and External Cues sessions will be video recorded to allow content to be tested in a lab study following the intervention. The research team worked with IT at STAR campus to position equipment so that the video only captures the interventionists (session leaders). Participants will not be recorded. If any participant audio is captured, content containing participants' voices will be deleted from the file. The purpose of recording is to modify the curriculum for future interventions and programs.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between the ages of 18 and 26
* Freshman, Sophomore, or Junior University of Delaware student
* Willing and able to commit to the 10-week study at the specified times and a follow up visit 1-year after the completion of the study
* Have concerns about body shape, weight, and/or eating
* Are not currently being treated for an eating disorder

Exclusion Criteria:

* They do not meet the inclusion criteria.
* They have a severe medical food allergy.
* They are pregnant - this program is not geared towards someone who is pregnant.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Intuitive Eating | Baseline - week 1
  Using the Intuitive Eating Scale-2 Measures tendency to follow physical hunger and fullness cues
  *Total*score range = 5-115 Higher scores indicate greater levels of intuitive eating or its dimensions
Intuitive Eating | Midpoint - week 5
  Using the Intuitive Eating Scale-2 Measures tendency to follow physical hunger and fullness cues
  *Total*score range = 5-115 Higher scores indicate greater levels of intuitive eating or its dimensions
Intuitive Eating | End of study - week 10
  Using the Intuitive Eating Scale-2 Measures tendency to follow physical hunger and fullness cues
  *Total*score range = 5-115 Higher scores indicate greater levels of intuitive eating or its dimensions
Intuitive Eating | Follow-up - 1 year post study completion
  Using the Intuitive Eating Scale-2 Measures tendency to follow physical hunger and fullness cues
  *Total*score range = 5-115 Higher scores indicate greater levels of intuitive eating or its dimensions
Interoceptive Awareness | Baseline - week 1
  Using the Multi-Dimensional Assessment of Interoceptive Awareness - 2 Measures the multiple levels of individual interoception
  *Total*score range = 0-185 Higher total scores and sub scale scores indicate higher levels of positive awareness
Interoceptive Awareness | Midpoint - week 5
  Using the Multi-Dimensional Assessment of Interoceptive Awareness - 2 Measures the multiple levels of individual interoception
  *Total*score range = 0-185 Higher total scores and sub scale scores indicate higher levels of positive awareness
Interoceptive Awareness | End of study - week 10
  Using the Multi-Dimensional Assessment of Interoceptive Awareness - 2 Measures the multiple levels of individual interoception
  *Total*score range = 0-185 Higher total scores and sub scale scores indicate higher levels of positive awareness
Interoceptive Awareness | Follow-up - 1 year post study completion
  Using the Multi-Dimensional Assessment of Interoceptive Awareness - 2 Measures the multiple levels of individual interoception
  *Total*score range = 0-185 Higher total scores and sub scale scores indicate higher levels of positive awareness
Dietary Restraint | Baseline - week 1
  Using the Three-Factor Eating Questionnaire-18 Measures dietary restraint Means are computed for three subscales and are transformed to a 0-100 scale score Higher scores indicate greater cognitive restraint, uncontrolled, emotional eating
Dietary Restraint | Midpoint - week 5
  Using the Three-Factor Eating Questionnaire-18 Measures dietary restraint Means are computed for three subscales and are transformed to a 0-100 scale score Higher scores indicate greater cognitive restraint, uncontrolled, emotional eating
Dietary Restraint | End of study - week 10
  Using the Three-Factor Eating Questionnaire-18 Measures dietary restraint Means are computed for three subscales and are transformed to a 0-100 scale score Higher scores indicate greater cognitive restraint, uncontrolled, emotional eating
Dietary Restraint | Follow-up - 1 year post study completion
  Using the Three-Factor Eating Questionnaire-18 Measures dietary restraint Means are computed for three subscales and are transformed to a 0-100 scale score Higher scores indicate greater cognitive restraint, uncontrolled, emotional eating
Embodiment | Baseline - week 1
  Using the Experience of Embodiment Scale - Body Connection and Comfort Subscale Measures one of the five dimensions of embodiment: body connection and comfort Subscale score range = 12-36 Higher sub scale scores indicate higher levels of embodiment in terms of connection and comfort to one's body
Embodiment | Midpoint - week 5
  Using the Experience of Embodiment Scale - Body Connection and Comfort Subscale Measures one of the five dimensions of embodiment: body connection and comfort Subscale score range = 12-36 Higher sub scale scores indicate higher levels of embodiment in terms of connection and comfort to one's body
Embodiment | End of study - week 10
  Using the Experience of Embodiment Scale - Body Connection and Comfort Subscale Measures one of the five dimensions of embodiment: body connection and comfort Subscale score range = 12-36 Higher sub scale scores indicate higher levels of embodiment in terms of connection and comfort to one's body
Embodiment | Follow-up - 1 year post study completion
  Using the Experience of Embodiment Scale - Body Connection and Comfort Subscale Measures one of the five dimensions of embodiment: body connection and comfort Subscale score range = 12-36 Higher sub scale scores indicate higher levels of embodiment in terms of connection and comfort to one's body
Body Appreciation | Baseline - week 1
  Using the Body Appreciation Scale - 2 Measures one's acceptance of, favorable opinions toward, and respect for their body Score answers are totaled and divided by 10 for an average score. *total* average scores can range from = 1-5 Higher scores indicate higher levels of body appreciation
Body Appreciation | Midpoint - week 5
  Using the Body Appreciation Scale - 2 Measures one's acceptance of, favorable opinions toward, and respect for their body Score answers are totaled and divided by 10 for an average score. *total* average scores can range from = 1-5 Higher scores indicate higher levels of body appreciation
Body Appreciation | End of study - week 10
  Using the Body Appreciation Scale - 2 Measures one's acceptance of, favorable opinions toward, and respect for their body Score answers are totaled and divided by 10 for an average score. *total* average scores can range from = 1-5 Higher scores indicate higher levels of body appreciation
Body Appreciation | Follow-up - 1 year post study completion
  Using the Body Appreciation Scale - 2 Measures one's acceptance of, favorable opinions toward, and respect for their body Score answers are totaled and divided by 10 for an average score. *total* average scores can range from = 1-5 Higher scores indicate higher levels of body appreciation

SECONDARY OUTCOMES:
Fruit Consumption | Baseline - week 1
  Using select modified questions from YRBS and Project EAT One question Measures fruit consumption in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many times did you eat fruit? (Do not count fruit juice).
  Score answers range from 1 to 7, with 1 being "I did not eat fruit during a typical week" and 7 being "4 or more times per day during a typical week" Higher scores indicate greater consumption of fruit in a typical week over the past 5 weeks
Fruit Consumption | Midpoint - week 5
  Using select modified questions from YRBS and Project EAT One question Measures fruit consumption in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many times did you eat fruit? (Do not count fruit juice).
  Score answers range from 1 to 7, with 1 being "I did not eat fruit during a typical week" and 7 being "4 or more times per day during a typical week" Higher scores indicate greater consumption of fruit in a typical week over the past 5 weeks
Fruit Consumption | End of study - week 10
  Using select modified questions from YRBS and Project EAT One question Measures fruit consumption in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many times did you eat fruit? (Do not count fruit juice).
  Score answers range from 1 to 7, with 1 being "I did not eat fruit during a typical week" and 7 being "4 or more times per day during a typical week" Higher scores indicate greater consumption of fruit in a typical week over the past 5 weeks
Fruit Consumption | Follow-up - 1 year post study completion
  Using select modified questions from YRBS and Project EAT One question Measures fruit consumption in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many times did you eat fruit? (Do not count fruit juice).
  Score answers range from 1 to 7, with 1 being "I did not eat fruit during a typical week" and 7 being "4 or more times per day during a typical week" Higher scores indicate greater consumption of fruit in a typical week over the past 5 weeks
Vegetable Consumption | Baseline - week 1
  Using select modified questions from YRBS and Project EAT One question Measures vegetable consumption in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many times did you eat vegetables? (Do not count green salad, potatoes, or carrots).
  Score answers range from 1 to 7, with 1 being "I did not eat vegetables during a typical week" and 7 being "4 or more times per day during a typical week" Higher scores indicate greater consumption of vegetables in a typical week over the past 5 weeks
Vegetable Consumption | Midpoint - week 5
  Using select modified questions from YRBS and Project EAT One question Measures vegetable consumption in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many times did you eat vegetables? (Do not count green salad, potatoes, or carrots).
  Score answers range from 1 to 7, with 1 being "I did not eat vegetables during a typical week" and 7 being "4 or more times per day during a typical week" Higher scores indicate greater consumption of vegetables in a typical week over the past 5 weeks
Vegetable Consumption | End of study - week 10
  Using select modified questions from YRBS and Project EAT One question Measures vegetable consumption in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many times did you eat vegetables? (Do not count green salad, potatoes, or carrots).
  Score answers range from 1 to 7, with 1 being "I did not eat vegetables during a typical week" and 7 being "4 or more times per day during a typical week" Higher scores indicate greater consumption of vegetables in a typical week over the past 5 weeks
Vegetable Consumption | Follow-up - 1 year post study completion
  Using select modified questions from YRBS and Project EAT One question Measures vegetable consumption in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many times did you eat vegetables? (Do not count green salad, potatoes, or carrots).
  Score answers range from 1 to 7, with 1 being "I did not eat vegetables during a typical week" and 7 being "4 or more times per day during a typical week" Higher scores indicate greater consumption of vegetables in a typical week over the past 5 weeks
Participation in Yoga | Baseline - week 1
  Using select modified questions from YRBS and Project EAT One question Measures participation in yoga in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many hours did you practice yoga?".
  Score answers range from 1 to 7, with 1 being "0 hours during a typical week" and 7 being "10+ hours during a typical week" Higher scores indicate greater frequency spent practicing yoga in a typical week over the past 5 weeks
Participation in Yoga | Midpoint - week 5
  Using select modified questions from YRBS and Project EAT One question Measures participation in yoga in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many hours did you practice yoga?".
  Score answers range from 1 to 7, with 1 being "0 hours during a typical week" and 7 being "10+ hours during a typical week" Higher scores indicate greater frequency spent practicing yoga in a typical week over the past 5 weeks
Participation in Yoga | End of study - week 10
  Using select modified questions from YRBS and Project EAT One question Measures participation in yoga in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many hours did you practice yoga?".
  Score answers range from 1 to 7, with 1 being "0 hours during a typical week" and 7 being "10+ hours during a typical week" Higher scores indicate greater frequency spent practicing yoga in a typical week over the past 5 weeks
Participation in Yoga | Follow-up - 1 year post study completion
  Using select modified questions from YRBS and Project EAT One question Measures participation in yoga in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many hours did you practice yoga?".
  Score answers range from 1 to 7, with 1 being "0 hours during a typical week" and 7 being "10+ hours during a typical week" Higher scores indicate greater frequency spent practicing yoga in a typical week over the past 5 weeks
Participation in Physical Activity | Baseline - week 1
  Using select modified questions from YRBS and Project EAT One question Measures participation in cardiovascular exercise in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many hours did you engage in cardio exercise? (Add up all the time you spent in any kind of physical activity that increased your heart rate and made you breathe hard some of the time)".
  Score answers range from 1 to 7, with 1 being "0 hours during a typical week" and 7 being "10+ hours during a typical week" Higher scores indicate greater frequency spent engaging in cardiovascular exercise in a typical week over the past 5 weeks
Participation in Physical Activity | Midpoint - week 5
  Using select modified questions from YRBS and Project EAT One question Measures participation in cardiovascular exercise in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many hours did you engage in cardio exercise? (Add up all the time you spent in any kind of physical activity that increased your heart rate and made you breathe hard some of the time)".
  Score answers range from 1 to 7, with 1 being "0 hours during a typical week" and 7 being "10+ hours during a typical week" Higher scores indicate greater frequency spent engaging in cardiovascular exercise in a typical week over the past 5 weeks
Participation in Physical Activity | End of study - week 10
  Using select modified questions from YRBS and Project EAT One question Measures participation in cardiovascular exercise in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many hours did you engage in cardio exercise? (Add up all the time you spent in any kind of physical activity that increased your heart rate and made you breathe hard some of the time)".
  Score answers range from 1 to 7, with 1 being "0 hours during a typical week" and 7 being "10+ hours during a typical week" Higher scores indicate greater frequency spent engaging in cardiovascular exercise in a typical week over the past 5 weeks
Participation in Physical Activity | Follow-up - 1 year post study completion
  Using select modified questions from YRBS and Project EAT One question Measures participation in cardiovascular exercise in a typical week over the past 5 weeks Question asks: "Thinking about the past 5 weeks, in a typical week, how many hours did you engage in cardio exercise? (Add up all the time you spent in any kind of physical activity that increased your heart rate and made you breathe hard some of the time)".
  Score answers range from 1 to 7, with 1 being "0 hours during a typical week" and 7 being "10+ hours during a typical week" Higher scores indicate greater frequency spent engaging in cardiovascular exercise in a typical week over the past 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carly Pacanowski, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No